CLINICAL TRIAL: NCT02557412
Title: Long-term Effect of Nasal Continuous Positive Airway Pressure on Lipid Profile in Patients With Dyslipidaemia and Mild-moderate Obstructive Sleep Apnea
Brief Title: Effect of Nasal CPAP on Lipid Profile in Patients With Dyslipidaemia and Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limitations to recruitment related to COVID
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario Principe de Asturias (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PINML01
Record Dates: First submitted 2015-06-25; First posted 2015-09-23 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Sleep Apnea; Dyslipidaemia
MeSH Terms: conditions — Sleep Apnea Syndromes; Dyslipidemias | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional treatment (Placebo Comparator): Hygiene and diet recommendations on sleep.
  Interventions: Other: Conventional treatment
- Intensive lifestyle intervention (Active Comparator): Lifestyle intervention will consist of a structured intervention in a specific alimentary plan (carbohydrates: 40-45%; fats: 25-35% [saturated fats <7% monounsaturated fats up to 20% and polyunsaturated fats <10% ] and proteins: 15-20%), which will be repeated in each review. Also, be recommended to increase daily physical activity, setting a target walking 10,000 steps a day. To do this, to patients assigned to this treatment arm, will be provided with a pedometer and will asked to fill out a form with the steps that they walked each day. At each visit, the distance walked will be reviewed and the target set will be remarked.
  Interventions: Behavioral: Intensive lifestyle intervention
- Continuous positive airway pressure (Active Comparator): Treatment with nasal continuous positive airway pressure (CPAP). Treatment begins with an empirical pressure of 8 centimetres of water (cmH2O) and in a period of three weeks, the pressure is adjusted by titration with an automatic positive airway pressure device (AutoSet II, ResMed).
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — Treatment with nasal CPAP. Treatment begins with an empirical pressure of 8 cmH2O and in a period of three weeks, the pressure is adjusted by automatic titration with AutoSet II (ResMed) device.
  Arms: Continuous positive airway pressure
Behavioral: Intensive lifestyle intervention — Specific alimentary plan (carbohydrates: 40-45%; fats: 25-35% [saturated fats <7% monounsaturated fats up to 20% and polyunsaturated fats <10% ] and proteins: 15-20%) and recommendation to increase daily physical activity, setting a target walking 10,000 steps a day. The patients will be provided with a pedometer and will asked to fill out a form with the steps that they walked each day. At each visit, the distance walked will be reviewed and the target set will be remarked.
  Arms: Intensive lifestyle intervention
Other: Conventional treatment — Hygiene and diet recommendations on sleep
  Arms: Conventional treatment

SUMMARY:
OBJECTIVES Main objective: To assess if six months of treatment with CPAP, associated with conventional treatment, improves the lipid profile of patients with dyslipidemia and mild-moderate apnea-hypopnea syndrome (OSA).

Secondary objectives:

* Determine the additional effect of CPAP on insulin resistance and dyslipidemia in patients with mild-moderate OSA.
* Assess the impact of CPAP treatment in reducing cardiovascular risk in patients with dyslipidemia and mild-moderate OSA.

DESIGN Randomized, parallel group, non-blind, controlled clinical trial with conventional treatment.

STUDY POPULATION 35-75 year old subjects, diagnosed with dyslipidemia in last six months and in stable treatment during the last month with diet, cholesterol lowering drug, and cholesterol LDL levels> 100 mg / dl in the last two successive visits clinics.

Sample size. 38 patients who completed the test in each treatment arm.

TREATMENT

Patients will be randomized to one of the following treatment arms form:

1. hygiene and dietary recommendations.
2. lifestyle intervention (more strict and promotion of daily physical activity and dietary control).
3. Treatment with positive airway pressure (CPAP).

ENDPOINTS:

Efficacy endpoints.

* Primary endpoint: LDL-cholesterol.
* Total cholesterol, HDL-cholesterol, triglycerides and C-reactive protein high sensitivity (hsCRP).
* Systemic Biomarkers: inflammatory (IL-6, IL-8 and tumor necrosis factor (TNF)-α), oxidative stress (8-isoprostane), endothelial damage (endothelin, vascular cell adhesion molecule 1 (VCAM-1) and Intercellular Adhesion Molecule 1 (ICAM-1)), sympathetic activity (neuropeptide Y) and appetite-regulating hormones (leptin, orexin A / hypocretin-1 and ghrelin).
* Fasting glucose, glycated hemoglobin (HbA1c), fasting insulin and Homeostasis Model Assessment (HOMA) index and quantitative insulin sensitivity check index (QUICKI), thyroid-stimulating hormone (TSH).
* Clinical questionnaires: short-form (SF)-12, EuroQoL, Functional Outcomes of Sleep Questionnaire (FOSQ) and International physical activity questionnaire (IPAQ).

Security endpoints.

* Notification of clinical adverse events.
* Compliance with CPAP (average hours use per day).
* Epworth Sleepiness Questionnaire.
* Development of cardiovascular events.

DETAILED DESCRIPTION:
OBJECTIVES

Main objective: To assess if six months of treatment with CPAP, associated with conventional treatment, improves the lipid profile of patients with dyslipidemia and mild-moderate apnea-hypopnea syndrome (OSA).

Secondary objectives:

* Determine the additional effect of CPAP on insulin resistance and dyslipidemia in patients with mild-moderate OSA.
* Assess the impact of CPAP treatment in reducing cardiovascular risk in patients with dyslipidemia and mild-moderate OSA.
* Analyze the impact of supplemental CPAP treatment on glycemic control and the concentration of hsCRP in patients with dyslipidemia and mild-moderate OSA.
* Establish the impact of supplemental CPAP treatment on quality of life related to health of patients with dyslipidemia and mild-moderate OSA.
* Evaluate the effect of CPAP on inflammatory cytokines, oxidative stress biomarkers, sympathetic tone and regulating hormones intake in patients with dyslipidemia and mild-moderate OSA.
* Correlate CPAP induced changes in lipid levels with the changes produced in the basal inflammatory response, oxidative stress, sympathetic activity and intake regulating hormones.
* Compare the effect of CPAP with promotion of daily physical activity on lipid profile in patients with dyslipidemia and mild-moderate OSA.
* Identify the subgroup of patients with uncontrolled dyslipidemia and mild-moderate OSA in wich six months of treatment with CPAP achieve a more pronounced reduction in blood lipids.

DESIGN Randomized, parallel group, non-blind, controlled clinical trial with conventional treatment.

STUDY POPULATION 35-75 year old subjects, diagnosed with dyslipidemia in last six months and in stable treatment during the last month with diet, cholesterol lowering drug, and cholesterol LDL levels> 100 mg / dl in the last two successive visits clinics.

Sample size. 38 patients who completed the test in each treatment arm.

TREATMENT

Patients will be randomized to one of the following treatment arms form:

1. hygiene and dietary recommendations.
2. lifestyle intervention (more strict and promotion of daily physical activity and dietary control).
3. Treatment with positive airway pressure (CPAP).

ENDPOINTS Efficacy endpoints.

* Primary endpoint: LDL-cholesterol.
* Total cholesterol, HDL-cholesterol, triglycerides and C-reactive protein high sensitivity (hsCRP).
* Systemic Biomarkers: inflammatory (IL-6, IL-8 and TNF-α), oxidative stress (8-isoprostane), endothelial damage (endothelin, VCAM-1 and ICAM-1), sympathetic activity (neuropeptide Y) and appetite-regulating hormones (leptin, orexin A / hypocretin-1 and ghrelin).
* Fasting glucose, glycated hemoglobin (HbA1c), fasting insulin and HOMA and QUICKI indexes, TSH.
* Clinical questionnaires: SF-12, EuroQoL, FOSQ and IPAQ.

Security endpoints.

* Notification of clinical adverse events.
* Compliance with CPAP (average hours use per day).
* Epworth Sleepiness Questionnaire.
* Development of cardiovascular events.

STATISTICAL PROCEDURES Data will be expressed as mean ± standard deviation, median (interquartile range) or percent, depending on type and distribution. For comparison between groups, or t-Student test, or the Mann-Whitney U-test or chi-square test will be used, as appropriate. The relationships between variables will be analyzed by Pearson correlation and multiple linear regression.

The treatment effect will be evaluated by analysis of variance for repeated measures with post-hoc multiple comparisons, using the Bonferroni test. A model of multiple logistic regression will be applied to determine the variables associated with treatment response. P values will be considered statistically significant <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dyslipidemia: The existence of a previous clinical diagnostic of dyslipidemia associated with lipid-lowering therapy. It is also considered patients who have an altered analytical, using the following cutoffs: total cholesterol ≥ 200 mg / dl, triglycerides ≥ 180 mg / dl, HDL-cholesterol ≤ 40 mg / dl or LDL-cholesterol ≥ 150 mg / dl. Lipid-lowering treatment and diet, stable in the last month.
* A concentration of LDL-cholesterol above 100 mg / dl, in the month prior to inclusion.
* An apnea-hypopnea index between 5-30 h-1

Exclusion Criteria:

* Apnea-hypopnea index of less than 5 h-1 or greater than 30 h-1.
* Predominance of central apneas and hypopneas, defined as more than 25% of all respiratory events.
* Professional drivers, risk profession or respiratory failure (according to criteria of the clinical pathway for diagnosis and treatment of sleep-disordered breathing).
* Very excessive daytime sleepiness (Epworth Sleepiness Scale> 18).
* Morbid obesity (BMI> 40 kg / m2).
* Prior treatment with CPAP.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol | 6 months
  LDL-cholesterol level in peripheral blood

SECONDARY OUTCOMES:
Lipid profile | 6 months
  Total cholesterol, HDL-cholesterol, and triglycerides
Systemic biomarkers | 6 months
  C-reactive protein, IL-6, IL-8, TNF-α, 8-isoprostane, endothelin, VCAM-1, ICAM-1, neuropeptide Y, leptin, orexin and ghrelin.
Glycated hemoglobin | 6 months
  Glycated hemoglobin (HbA1c).
Insulin resistance | 6 months
  HOMA and QUICKI indexes.
Health-related quality of life | 6 months
  SF-12, EuroQoL and FOSQ questionnaires (generic and specific health-related quality of life).
Daily physical activity | 6 months
  IPAQ questionnaire.
Clinical adverse events | 6 months
CPAP compliance | 6 months
  Mean of CPAP use per night (h/night)
Sleepiness | 6 months
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, MD, Study Director — Hospital Universitario La Paz, IdiPAZ
Locations (1):
- Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid, Spain